CLINICAL TRIAL: NCT06065280
Title: Sodium-glucose Transport 2 Inhibitors (SGLT2i) in Heart Failure Reduced Ejection Fraction (HFrEF) Patients
Brief Title: Sodium-glucose Transport 2 Inhibitors (SGLT2i) in HFrEF Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Associate Professor, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SGLT2i in Heart Failure
Record Dates: First submitted 2023-09-27; First posted 2023-10-03 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure; Reduced Ejection Fraction Heart Failure
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic | interventions — empagliflozin; dapagliflozin

STUDY DESIGN:
Intervention Model Description: 80 patients with established heart failure reduced ejection fraction on optimal standard medical therapy, who will be consecutively randomly allocated to the SGLT2i (10 mg once a day Empagliflozin or Dapagliflozin ) with 40 patients with diabetes mellitus group and 40 patients non-diabetes mellitus group. (Each group will be divided into 2 subgroups one on Empagliflozin and the other one on Dapagliflozin )
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetic/HFrEF Group (Experimental): 40 patients with diabetes mellitus patients will be divided into 2 subgroups one on Empagliflozin and the other one on Dapagliflozin.
  Interventions: Drug: Empagliflozin 10 MG; Drug: Dapagliflozin 10 MG
- Nondiabetic/HFrEF Group (Experimental): 40 patients non-diabetes mellitus group will be divided into 2 subgroups one on Empagliflozin and the other one on Dapagliflozin.
  Interventions: Drug: Empagliflozin 10 MG; Drug: Dapagliflozin 10 MG

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Each group will be divided into 2 subgroups one on Empagliflozin and the other one on Dapagliflozin 10 MG daily.
  Other Names: Jardiance 10 mg
Drug: Dapagliflozin 10 MG — Each group will be divided into 2 subgroups one on Empagliflozin and the other one on Dapagliflozin 10 MG daily.
  Other Names: Forxiga 10 mg

SUMMARY:
The aim of this study is to assess the efficacy, safety and cardiovascular outcomes of Sodium-glucose transport protein 2 inhibitors (SGLT2i) therapy in patients with heart failure reduced ejection fraction ( HFrEF) with and without diabetes mellitus and is to evaluate short-term effect of these drugs using the cardiac biomarkers Neopterin.

DETAILED DESCRIPTION:
* A 3 months, prospective interventional study, which will include 80 patients with established heart failure reduced ejection fraction on optimal standard medical therapy, who will be consecutively randomly allocated to the SGLT2i (10 mg once a day Empagliflozin or Dapagliflozin ) with 40 patients with diabetes mellitus group and 40 patients non-diabetes mellitus group. (Each group will be divided into 2 subgroups one on Empagliflozin and the other one on Dapagliflozin )
* Approval will be obtained from Research Ethics Committee of Faculty of Pharmacy, Damanhour University

All patients will undergo :

* Provided written informed consent and entered a 10-day screening period, during which the trial inclusion and exclusion criteria were checked and baseline information gathered.
* Complete history with NYHA class assessment and clinical examination before and after the study
* 12-lead ECG before and after the study
* Complete Echocardiography study before and after the study
* Baseline venous sampling for urea, creatinine, potassium ,CBC , fasting blood sugar and Hemoglobin A1C at the beginning of the study and after 3 months of the study
* Measurements of Neopterin by ELISA at the beginning of the of the study and after 3 months of the study

Outcomes :

* Clinical outcomes, all patients will be followed up for 3 months for:
* 1ry outcomes: A)Complete Echocardiography monitoring for improvements B) Level of Neopterin C)will be a composite of worsening heart failure requiring hospitalization and/ or death from cardiovascular causes.
* 2ry outcomes: A) will be the additional secondary outcomes were the total number of hospitalizations for heart failure B) functional capacity and quality of life by the Kansas City Cardiomyopathy Questionnaire (KCCQ) reflects key health status.

C) a composite of worsening renal function, which will defined as a sustained decline in the eGFR of 50% or greater, end-stage renal disease (defined as a sustained [≥28 days] eGFR of <15 ml per minute per 1.73 m2, sustained dialysis, or renal transplantation), or renal death; and death from any cause.

• Safety outcomes : included serious adverse events, adverse events associated with the discontinuation of a trial treatment, adverse events of interest (i.e., volume depletion, renal events, major hypoglycemic events, diabetic ketoacidosis, dizziness , syncope ,acute renal failure or dialysis and laboratory findings of note, hypoglycemia and hypokalemia

ELIGIBILITY:
Inclusion criteria:

* Patients with HFrEF, on optimal medical therapy according to European Society of Cardiology guidelines,
* an age of at least 18 years,
* an ejection fraction of 40% or less, with New York Heart Association (NYHA) class II - IV symptoms will be eligible for the study.

Exclusion criteria:

* Recent treatment with or unacceptable side effects associated with an SGLT2i
* Type-I diabetes mellitus,
* Symptoms of hypotension or a systolic blood pressure of less than 95 mm Hg,
* Severe CKD and an estimated glomerular filtration rate (eGFR) below 30 ml per minute per 1.73 m2 of body-surface area or rapidly declining renal function
* Inability to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Neopterin Concentration | 3 month
  Neopterin serum level pg/ml

SECONDARY OUTCOMES:
hospitalization rate | 3 month
  hospitalizations duration (days)

CONTACTS AND LOCATIONS:
Overall Officials: Rehab H Werida, Ass Prof., Study Chair — Damanhour University
Locations (1):
- Damanhour Teaching Hospital, General Organization for Teaching Hospitals and Institutes., Damanhūr, Elbehairah, Egypt